CLINICAL TRIAL: NCT05955001
Title: A Randomized Controlled Trial to Examine the Utility of Tadalafil (5mg) For Treatment of Early Storage Symptoms and Erectile Dysfunction After Anatomical Endoscopic Enucleation of Prostate (AEEP)
Brief Title: Efficacy of Tadalafil (5mg) For Treatment of Early Storage Symptoms and Erectile Dysfunction After Endoscopic Enucleation of Prostate
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Laymon, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS.22.11.2208
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Erectile Dysfunction; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Erectile Dysfunction; Lower Urinary Tract Symptoms | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil 5 mg daily (Experimental): those patients will receive Tadalafil 5 mg daily after HoLEP
  Interventions: Drug: Tadalafil 5mg / Placebo
- Placebo (Experimental): Those patients will receive Placebo after HoLEP
  Interventions: Drug: Tadalafil 5mg / Placebo

INTERVENTIONS:
Drug: Tadalafil 5mg / Placebo — Patients after Holmium laser Enucleation of Prostate (HoLEP) will receive single daily dose of Tadalafil for 3 months and compared to Placebo
  Other Names: Placebo

SUMMARY:
From previous studies, the investigators found that sexual outcomes after prostate surgery may show insignificant improvement, remain unchanged or deteriorate in non-negligible number of patients especially those with high preoperative IIEF scores. Deterioration of erectile function could be attributed to persistence of storage symptoms specially nocturia. Several pathophysiologic mechanisms, described before, are involved in pathogenesis of LUTS and ED and one can imagine that after relief of obstruction, the erectile function should improve, however lack of improvement or even deterioration suggests that damage associated with these mechanisms is irreversible and patients may require some sort of penile rehabilitation after surgery.

The investigators hypothesized that Tadalafil may enhance relief of storage symptoms and enhance recovery of erectile function after surgery for BPH. With this assumption, a RCT was designed to examine the utility and efficacy of Tadalafil, once daily dose, to relieve persistent/ de novo storage symptoms and early erectile function deterioration after endoscopic prostate surgery.

DETAILED DESCRIPTION:
I. Introduction

Benign prostatic hyperplasia (BPH) accompanied by bothersome lower urinary tract symptoms (LUTS) is a common and progressive condition that significantly affects quality of life (QOL) in men. LUTS include storage, voiding, and post-micturition symptoms. Storage symptoms are referred as particularly bothersome and cause significant morbidity . Several population based studies demonstrated a strong association between LUTS and erectile dysfunction (ED) among BPH patients. This is believed to be independent of age and associated comorbidities like cardiovascular disease and diabetes mellitus.

Several mechanisms have been postulated to explain the relationship between LUTS and ED. First, impairment of nitric oxide (NO) production specially with conditions like hypertension and metabolic syndrome . Second, enhanced Rho/ROCK pathway that leads to impaired smooth muscle relaxation resulting in ED and LUTS. Overexpression of Rho/ROCK pathway has been found in hypertensive rats . Third, sympathetic over- activity, in particular, overexpression of α1A and α1D adrenergic receptors that are present mainly in prostate and hypertrophied detrusor muscle, respectively. Experimental studies demonstrated that hypertensive rats had increased sympathetic innervation to bladder and prostate, LUTS and ED. Furthermore, improvement of ED occurred after control of hypertension. Lastly, pelvic ischemia that results from atherosclerosis plays an important role in development of LUTS and ED via induction of fibrosis and decreased NO levels. In a cross sectional study by Berger et al , the authors found that patients with BPH and ED had lower perfusion and higher resistive index of the transition zone of prostate compared to young adults.

The main objective for treatment of BPH is to relieve LUTS and consequently improving quality of life. Anatomical endoscopic enucleation of prostate (AEEP) including, HoLEP and ThuLEP is recommended by the European Urological Association guideline as an efficient and advanced minimally invasive, size-independent surgical therapy of BPO. Their long-term efficacy, durability and safety have been proven in several prospective and randomized controlled studies .

I.1 Problems frequently encountered after AEEP that affect quality of life.

I.1.1 Persistent or De novo Storage Symptoms

Following HoLEP, a significant proportion of patients complain of persistent or even de novo storage symptoms. In a randomized trial comparing between HoLEP and TURP, Montorsi et al found that 44% of HoLEP patients experienced urgency, dysuria and urgency incontinence. Ahyai and colleagues prospectively analysed the incidence of storage symptoms after HoLEP among 144 patients. They found a significant (rebound) increase in storage symptoms at 6th and 8th week postoperatively that was attributed to the wound healing process and tissue edema. Moreover, persistence of storage symptoms led to delayed improvement in QoL that didn't significantly improved till 12 weeks after surgery when storage symptoms subsided.

Elkoushy et al compared the incidence of postoperative storage symptoms between HoLEP and PVP and found a significantly lower incidence in HoLEP group . The authors identified, baseline IPSS-storage subscore≥9, prolonged operative time>100 minutes and lower percentage of postoperative PSA reduction as independent predictors of less improvement of postoperative storage symptoms.

I.1.2. Sexual function deterioration

The impact of HoLEP on sexual function has been extensively addressed in literature with conflicting results. Some studies showed that HoLEP resulted in reduction of International Index of Erectile Function (IIEF) questionnaires postoperatively because of retrograde ejaculation that lowered IIEF orgasmic function domain . In a prospective controlled study, Elshal et al demonstrated a decline in erectile function (EF) domain after HoLEP in patients with normal preoperative EF (score >25). The authors also noted higher utilization of PDE5I from 27% to 30% at last follow up . In a retrospective study comparing effects of HoLEP, HoLAP and PVP on sexual function, the authors reported a decline in IIEF in 17% of patients after HoLEP . Higher baseline IIEF and high Energy/Prostate ratio were independent predictors of sexual function deterioration. In a recent prospective study including 144 patients treated with HoLEP, significant deterioration of IIEF for 24 weeks follow up after surgery. Jeong et al analysed serial changes in sexual function at 1,3,6 and 12 months after HoLEP and found early deterioration and return to baseline at 12 months follow up.

Theoretically, HoLEP has minimal effects on erection because of its pulsed nature, shallow depth of penetration (0.4mm) and majority of the procedure is performed with bunt dissection and laser energy is used mainly for control of blood vessels. Thus, the potential thermal effect on cavernous tissue or neurovascular bundles is minimal. Other factors could be attributed to early decline in erectile function including: anxiety after surgery, pain, postoperative complications, lack of ejaculation and bothering LUTS. Kim et al evaluated sexual outcomes after HoLEP using MSHQ and found a strong correlation between postoperative erectile function and nocturia. The authors explained their finding as decrease in nocturia led to better sleep quality and decreased overall physical fatigue thus increasing penile tumescence and erections.

I.2. Can penile rehabilitation enhance recovery of erectile function??? The concepts of penile rehabilitation has been studied after radical prostatectomy (RP) and can be defined as the use of any drug or device at or after RP to maximize erectile function recovery. Although there are different treatment methods used in penile rehabilitation, the most common approach of penile rehabilitation after RP are oral phosphodiesterase type 5 inhibitors (PDE5-I). Tadalafil is a long-acting PDE5 inhibitor (PDE5-I) that has been approved by US Food and Drug Administration (FDA) and by the European Medical Agency (EMA) for men with BPH-LUTS and for those with coexisting erectile dysfunction (ED) and BPH-LUTS. Clinical studies showed that Tadalafil improved symptoms of BPH, including both storage and voiding symptoms, in men with or without erectile dysfunction (ED).

I.3. Role of Phosphodiesterase 5 inhibitors (PDE5Is) in treatment of LUTS/ED

Mechanism of action:

PDE5 isoenzymes are highly expressed in human lower urinary tract (LUT) tissues. PDE5Is increase intracellular cyclic guanosine monophosphate (cGMP), leading to smooth muscle relaxation. The effect of PDE5 inhibition leading to elevated NO/cGMP concentration in the corpus cavernosum and pulmonary arteries has been observed, as well, in the smooth muscle of the prostate and bladder and their vascular supply. Moreover, chronic treatment with PDE5Is seems to increase blood perfusion and oxygenation in the LUT reducing chronic pelvic ischemia with its related functional and morphologic changes on bladder and prostate. PDE5I could also reduce chronic inflammation in the prostate and bladder. Nitric oxide and PDE5Is might also alter reflex pathways in the spinal cord and neurotransmission in the urethra, prostate, or bladder decreasing perception of bladder fullness and feeling of urgency.

II. Aim of the work From previous studies, we can conclude that sexual outcomes after prostate surgery may show insignificant improvement, remain unchanged or deteriorate in non-negligible number of patients especially those with high preoperative IIEF scores. Deterioration of erectile function could be attributed to persistence of storage symptoms specially nocturia. Several pathophysiologic mechanisms, described before, are involved in pathogenesis of LUTS and ED and one can imagine that after relief of obstruction, the erectile function should improve, however lack of improvement or even deterioration suggests that damage associated with these mechanisms is irreversible and patients may require some sort of penile rehabilitation after surgery.

The investigators hypothesized that Tadalafil may enhance relief of storage symptoms and enhance recovery of erectile function after surgery for BPH. With this assumption, a RCT was designed to examine the utility and efficacy of Tadalafil, once daily dose, to relieve persistent/ de novo storage symptoms and early erectile function deterioration after endoscopic prostate surgery.

Update (June 2025):

The initially listed time frame for outcome measures as "6 months" was a typographical error during registration. In practice, patients received Tadalafil or placebo for 3 months, and the primary assessment of orgasm perception (IIEF-15 domain) was conducted at 1 and 3 months while the patient was on treatment. The 6-month assessment represents post-treatment follow-up to evaluate symptom durability and resolution of postoperative recovery factors. No changes were made to outcome definitions or study design.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥ 40 years
* LUTS secondary to BOO due to BPH who failed medical treatment
* International prostate symptom scores (IPSS) >15 and bother score (QOL) ≥ 3 (according to IPSS question 8)
* Peak urinary flow rate (Qmax) <15 ml/sec.
* ASA (American society of anaesthesiologists) score ≤ 3.
* Sexually active men, not receiving PDE5I

Exclusion Criteria:

* Patients using nitrates, potassium channel opener, or α1-blockers doxazosin and terazosin for control of hypertension
* Patients with unstable angina pectoris, recent myocardial infarction or stroke myocardial insufficiency.
* Patients with severe hepatic or renal insufficiency.
* Patients who are sexually inactive.
* Patients with uncontrolled diabetes mellitus or neurologic condition(eg. parkinsoism)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Orgasm perception domain of International Index of Erectile Function (IIEF-15) questionnaire at 6 months among the study groups | 1 and 3 months postoperatively (during treatment), and at 6 months postoperatively (3 months after treatment cessation)
  the erectile function will be assessed using a validated questionnaire and compared to baseline .

SECONDARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) with its subdomains voiding and storage once at different follow up points. | 2 weeks, 1, 3 months (during treatment) and at 6 months postoperatively ( 3 months after treatment cessation)
  patients in the experimental group will also be evaluated in terms of urinary symptoms and whether their irritative symptoms were improved in comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Laymon, MD,MRCS, Principal Investigator — Urology and nephrology center, Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided